CLINICAL TRIAL: NCT00542815
Title: A Phase III, Multicentre, Open Label, Flexible Dose, Long Term Safety Study of MCI-196 in Chronic Kidney Disease Stage V Subjects on Dialysis With Hyperphosphatemia
Brief Title: A Study of MCI-196 in Chronic Kidney Disease Stage V Subjects on Dialysis With Hyperphosphatemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCI-196-E10
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Results first posted 2014-09-23 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Dialysis; Hyperphosphatemia
Keywords: Chronic Kidney Disease; Dialysis; Hyperphosphatemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — cholebine; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MCI-196
- 2 (Active Comparator)
  Interventions: Drug: Another Phosphate binder (Sevelamer)

INTERVENTIONS:
Drug: MCI-196 — 3g to 15g/day (3 times a day), Tablet, 40 weeks of flexible dose
  Other Names: Colestilan(INN); Colestimide(JAN); CHOLEBINE®; BindRen®
  Arms: 1
Drug: Another Phosphate binder (Sevelamer) — Current approved dosing recommendations for 12 weeks
  Arms: 2

SUMMARY:
This is a PIII multi-center, open-label, flexible dose, long-term safety study, that in conjunction with the E07(NCT00416520), E08(NCT00542386) and E09(NCT00451295) studies will allow exposure to MCI-196 for up to 52 weeks

DETAILED DESCRIPTION:
Following completion of one of the Phase III studies (E07, E08 or E09) eligible patients will receive either MCI-196 for up to 52 weeks. The study is in two periods. The initial period allows flexible dosing for a period of 8 weeks. This will allow subjects to achieve individually optimised doses. After 8 weeks, subjects will continue flexible dosing with MCI-196 but with titration intervals every 4 weeks instead of every 2 weeks. Subjects previously exposed to MCI-196 will end the study at Week 40.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable haemodialysis or peritoneal dialysis treatment.
* Stable phosphate control
* Stabilised phosphorus diet.
* female subjects of child-bearing potential must have a negative serum pregnancy test.
* Male subjects must agree to use appropriate contraception.
* Completed one of the MCI-196 PIII studies

Exclusion Criteria:

* Current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose them to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* Body Mass Index (BMI) <= 16.0 kg/m2 or =>40.0 kg/m2.
* Current or a history of significant gastrointestinal motility problems
* Positive test for HIV 1 and 2 antibodies.
* History of substance or alcohol abuse within the last year.
* Seizure disorders.
* History of drug or other allergy.
* Temporary catheter with active signs of inflammation or infection.
* The subject has participated in a clinical study with any experimental medication (with the exception of MCI-196 PIII studies) in the last 30days or experimental biological product within the 90 days prior to signing of informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2007-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma Europe
Locations (115):
- Graz, Austria
- Czechia (6):
  - Frýdek-Místek
  - Hradec Králové
  - Ostrava
  - Prague
  - Tábor
  - Ústí nad Labem
- France (3):
  - Bordeaux
  - Montpelier
  - Paris
- Germany (9):
  - Aschaffenburg
  - Coesfeld
  - Darmstadt
  - Dortmund
  - Düsseldorf
  - Hamburg
  - Homberg (Efze)
  - Langen
  - Mannheim-Kafertal
- Hungary (8):
  - Ajka
  - Baja
  - Budapest
  - Esztergom
  - Győr
  - Hatvan
  - Kisvárda
  - Veszprém
- Italy (12):
  - Ancona
  - Cernusco sul Naviglio
  - Como
  - Cremona
  - Lecco
  - Livorno
  - Milan
  - Modena
  - Ostia Roma
  - Pavia
  - Perugia
  - Rome
- Malaysia (9):
  - Alor Star
  - Klang
  - Kota Kinabalu
  - Kuala Terengganu
  - Kuching
  - Malacca
  - Selangor Darul Ehsan
  - Seremban
  - Taiping
- Skopje, North Macedonia
- Poland (16):
  - Ciechanów
  - Częstochowa
  - Gdansk
  - Lodz
  - Lublin
  - Oświęcim
  - Pabianice
  - Poznan
  - Rybnik
  - Sokołów Podlaski
  - Starogard Gdański
  - Warsaw
  - Wejherowo
  - Wroclaw
  - Zgierz
  - Zielona Góra
- Russia (26):
  - Arkhangelsk
  - Chita
  - Irkutsk
  - Ivanovo
  - Kaluga
  - Karbysheva str.Volzskiy
  - Kemerovo
  - Khabarovsk
  - Krasnodar
  - Krasnoyarsk
  - Moscow
  - Mytishchi
  - Nizhny Novgorod
  - Novokuznetsk
  - Novorossiysk
  - Novosibirsk
  - Omsk
  - Petrozavodsk
  - Rostov-on-Don
  - Rozhkova
  - Saint Petersburg
  - Smolensk
  - Tomsk
  - Vladivostok
  - Yaroslavl
  - Yekaterinburg
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
- South Africa (5):
  - Cape Town
  - Durban
  - Gauteng
  - Johannesburg
  - Port Elizabeth
- Spain (3):
  - Barcelona
  - Oviedo
  - Seville
- Ukraine (10):
  - Chernivtsy
  - Dnipro
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Mykolayiv
  - Ternopil
  - Uzhhorod
  - Zaporizhya
  - Zhytomyr
- United Kingdom (2):
  - Glasgow
  - Stevenage

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-196 From E07 / E08 Studies; MCI-196 From E07 Study: 3, 6, 9, 12, or 15g / day as titrated
- Sevelamer From E07 Study: 2.4, 4.8, 7.2, 9.6, or 12.0g / day as titrated
Period: Overall Study
Arm/Group | MCI-196 From E07 / E08 Studies | MCI-196 From E07 Study | Sevelamer From E07 Study
Started | 432 | 76 | 124
Completed | 326 | 44 | 92
Not Completed | 106 | 32 | 32
Not completed — Adverse Event | 19 | 6 | 9
Not completed — Death | 10 | 7 | 3
Not completed — Lack of Efficacy | 9 | 2 | 0
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Withdrawal by Subject | 41 | 5 | 8
Not completed — Other reasons | 24 | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-196 From E07 / E08 Studies | MCI-196 From E07 Study | Sevelamer From E07 Study | Total
Number analyzed (Participants) | 432 | 76 | 124 | 632
Age, Customized [Number; unit: participants]
  <65 years | 374 | 55 | 77 | 506
  >=65 years | 58 | 21 | 47 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 25 | 53 | 281
  Male | 229 | 51 | 71 | 351

OUTCOME MEASURES:

1. Primary Outcome: The Change in Serum Phosphorus for MCI-196 and Sevelamer
Description: Change from Baseline to Week 52 (LOCF)
Time Frame: 52 weeks (Baseline-52 weeks)
Population: ITT2 population included all subjects who received enrolment number into MCI-196-E10, took at least 1 dose of study medication in original study and had at least 1 post-enrolment efficacy value after start of study medication in MCI-196-E10. Data collected from start of original studies to end of MCI-196-E10 were analysed for this population.
Measure: Mean (Standard Deviation); unit: mg / dL
Arm/Group | MCI-196 From E07 / E08 Studies | MCI-196 From E07 Study | Sevelamer From E07 Study
Number analyzed (Participants) | 429 | 75 | 124
mg / dL | -1.23 (1.78) | -1.47 (1.68) | -2.26 (1.82)

2. Secondary Outcome: The Percent Change in Serum LDL-cholesterol for MCI-196 and Sevelamer
Description: Percent Change from Baseline to Week 52 (LOCF)
Time Frame: 52 weeks (Baseline-52 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change of LDL-cholesterol
Arm/Group | MCI-196 From E07 / E08 Studies | MCI-196 From E07 Study | Sevelamer From E07 Study
Number analyzed (Participants) | 429 | 75 | 124
percentage change of LDL-cholesterol | -26.22 (27.08) | -30.62 (20.12) | -28.66 (23.61)

ADVERSE EVENTS:
Groups:
- MCI-196 From E07/E08 Studies; MCI-196 From E07 Study: 3, 6, 9, 12, or 15g / day as titrated
Arm/Group | MCI-196 From E07/E08 Studies | MCI-196 From E07 Study | Sevelamer From E07 Study
Serious Adverse Events (participants affected / at risk) | 74/432 | 31/76 | 48/124
Other Adverse Events (participants affected / at risk) | 310/432 | 75/76 | 112/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 From E07/E08 Studies (N=432) | MCI-196 From E07 Study (N=76) | Sevelamer From E07 Study (N=124)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 3 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Parathyroid gland enlargement (Endocrine disorders) | 1 | 1 | 0
Iritis (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 3 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Cardiac death (General disorders) | 1 | 1 | 0
Catheter related complication (General disorders) | 1 | 0 | 0
Catheter site haematoma (General disorders) | 1 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Catheter site phlebitis (General disorders) | 1 | 0 | 0
Mass (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Aeromona infection (Infections and infestations) | 1 | 1 | 0
Arteriovenous fistula site infection (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Catheter sepsis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 7 | 3 | 1
Pyelonephritis chronic (Infections and infestations) | 1 | 0 | 0
Pyonephrosis (Infections and infestations) | 1 | 1 | 0
Salpingitis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Wound sepsis (Infections and infestations) | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 2 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 5 | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dialysis device complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Shunt malfunction (Injury, poisoning and procedural complications) | 1 | 1 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arteriogram coronary (Investigations) | 1 | 1 | 2
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 1 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Encephalomalacia (Nervous system disorders) | 1 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 2
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0
Reduced bladder capacity (Renal and urinary disorders) | 1 | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Arteriosclerosis obliterans (Vascular disorders) | 1 | 1 | 0
Brachiocephalic vein stenosis (Vascular disorders) | 2 | 2 | 1
Circulatory collapse (Vascular disorders) | 2 | 2 | 0
Extremity necrosis (Vascular disorders) | 1 | 1 | 2
Haematoma (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0 | 3
Hypovolaemic shock (Vascular disorders) | 1 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1
Venous insufficiency (Vascular disorders) | 1 | 0 | 0
Venous occlusion (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 From E07/E08 Studies (N=432) | MCI-196 From E07 Study (N=76) | Sevelamer From E07 Study (N=124)
Anaemia (Blood and lymphatic system disorders) | 34 | 13 | 22
Nephrogenic anaemia (Blood and lymphatic system disorders) | 6 | 2 | 1
Angina pectoris (Cardiac disorders) | 5 | 1 | 4
Myocardial ischaemia (Cardiac disorders) | 9 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 6 | 1 | 4
Hyperparathyroidism (Endocrine disorders) | 14 | 5 | 12
Hyperparathyroidism secondary (Endocrine disorders) | 5 | 3 | 4
Conjunctivitis (Eye disorders) | 6 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 14 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 21 | 9 | 13
Abdominal pain upper (Gastrointestinal disorders) | 25 | 8 | 7
Constipation (Gastrointestinal disorders) | 32 | 14 | 14
Diarrhoea (Gastrointestinal disorders) | 31 | 15 | 20
Duodenitis (Gastrointestinal disorders) | 4 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 40 | 13 | 9
Flatulence (Gastrointestinal disorders) | 9 | 2 | 3
Gastritis (Gastrointestinal disorders) | 10 | 3 | 2
Gastritis erosive (Gastrointestinal disorders) | 9 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 50 | 8 | 13
Oesophagitis (Gastrointestinal disorders) | 3 | 3 | 1
Toothache (Gastrointestinal disorders) | 3 | 3 | 3
Vomiting (Gastrointestinal disorders) | 37 | 15 | 13
Asthenia (General disorders) | 19 | 3 | 2
Non-cardiac chest pain (General disorders) | 4 | 2 | 2
Oedema peripheral (General disorders) | 16 | 9 | 4
Pyrexia (General disorders) | 12 | 2 | 7
Bronchitis (Infections and infestations) | 15 | 8 | 11
Catheter sepsis (Infections and infestations) | 2 | 2 | 1
Cystitis (Infections and infestations) | 3 | 0 | 5
Gastroenteritis (Infections and infestations) | 2 | 0 | 3
Influenza (Infections and infestations) | 13 | 3 | 8
Nasopharyngitis (Infections and infestations) | 13 | 8 | 14
Pharyngitis (Infections and infestations) | 7 | 3 | 5
Respiratory tract infection (Infections and infestations) | 10 | 4 | 0
Respiratory tract infection viral (Infections and infestations) | 9 | 0 | 0
Rhinitis (Infections and infestations) | 5 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 8
Urinary tract infection (Infections and infestations) | 5 | 3 | 6
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 7 | 6 | 2
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 5
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 13 | 3 | 5
Dialysis device complication (Injury, poisoning and procedural complications) | 3 | 2 | 1
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 22 | 8 | 13
Limb injury (Injury, poisoning and procedural complications) | 1 | 1 | 3
Procedural hypertension (Injury, poisoning and procedural complications) | 14 | 2 | 6
Procedural hypotension (Injury, poisoning and procedural complications) | 16 | 6 | 9
Procedural pain (Injury, poisoning and procedural complications) | 3 | 3 | 1
Blood parathyroid hormone increased (Investigations) | 14 | 2 | 7
C-reactive protein increased (Investigations) | 5 | 5 | 7
Electrocardiogram QT interval abnormal (Investigations) | 2 | 2 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 13 | 4 | 3
Fluid overload (Metabolism and nutrition disorders) | 2 | 2 | 3
Fluid retention (Metabolism and nutrition disorders) | 8 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 6 | 7
Hyperphosphataemia (Metabolism and nutrition disorders) | 7 | 3 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 32 | 12 | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Iron deficiency (Metabolism and nutrition disorders) | 2 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 3 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 10 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 13 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3 | 13
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Headache (Nervous system disorders) | 31 | 9 | 12
Anxiety (Psychiatric disorders) | 5 | 3 | 2
Insomnia (Psychiatric disorders) | 6 | 1 | 4
Anuria (Renal and urinary disorders) | 2 | 2 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 8 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 6 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Renal transplant (Surgical and medical procedures) | 12 | 7 | 5
Accelerated hypertension (Vascular disorders) | 2 | 2 | 1
Arteriosclerosis (Vascular disorders) | 2 | 1 | 3
Hypertension (Vascular disorders) | 55 | 23 | 39
Hypotension (Vascular disorders) | 13 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other